CLINICAL TRIAL: NCT01959958
Title: Evaluation of Nocturnal Enuresis and Barriers to Treatment Among Pediatric Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PEESC
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Sickle Cell Disease
Keywords: Nocturnal enuresis; Barriers to treatment
MeSH Terms: conditions — Anemia, Sickle Cell; Nocturnal Enuresis | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle cell disease: In this study, children and adolescents with sickle cell disease ages 6-18 years and their parents/guardians will complete a questionnaire/interview.
  Interventions: Other: Questionnaire/Interview

INTERVENTIONS:
Other: Questionnaire/Interview — Participants will each complete an interview with questionnaires assessing nocturnal enuresis, health-related quality of life, emotional and behavioral functioning, family functioning, and stressful life events. Participants who report nocturnal enuresis will also be asked to identify interventions they have used in the past, along with barriers to intervention implementation.

SUMMARY:
Pediatric patients with sickle cell disease are at greater risk for exhibiting nocturnal enuresis (bedwetting) compared to the general population. This increased risk has been attributed to a decreased ability to concentrate urine caused by sickling-induced nephropathy. The sociodemographic, psychosocial, and medical factors associated with nocturnal enuresis are not well defined. In addition, the impact of these behaviors on emotional and behavioral functioning, along with health-related quality of life are not clear. Despite the availability of evidence-based interventions for nocturnal enuresis, very few families with a child with sickle cell disease have utilized these methods. The reasons for this underutilization of interventions are not clear.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: To examine differences between those who do and those who do not exhibit nocturnal enuresis in regard to health-related quality of life, emotional and behavioral functioning, family functioning, stressful life events, sociodemographic factors and medical factors.

SECONDARY OBJECTIVE: To identify barriers to intervention implementation for nocturnal enuresis.

In this study, children and adolescents with sickle cell disease ages 6-18 years and their parents/guardians will each complete an interview with questionnaires assessing nocturnal enuresis, health-related quality of life, emotional and behavioral functioning, family functioning, and stressful life events. Participants who report nocturnal enuresis will identify interventions they have used in the past, along with barriers to intervention implementation.

The future goal will be to use this information to develop an effective intervention strategy for nocturnal enuresis specific to the needs of children and adolescents with sickle cell disease.

ELIGIBILITY:
INCLUSION CHARACTERISTICS:

* Child Characteristics:

  * St. Jude Children's Research Hospital (SJCRH) patient with a primary diagnosis of sickle cell disease (HbSS, HbSC, HbSβ0thalassemia, HbSβ+thalassemia)
  * Age 6.0-17.99 years at the time of enrollment
  * Primary language is English
  * Has the cognitive capacity to complete questionnaires
* Caregiver Characteristics:

  * Parent or guardian of SJCRH patient who meets above criteria
  * Primary language is English
  * Has the cognitive capacity to complete questionnaires

EXCLUSION CRITERIA:

* Child Characteristics:

  * Experiencing current acute complications of sickle cell disease requiring hospitalization or an acute care visit (e.g., pain crises, acute chest syndrome, acute cerebrovascular events/stroke or active infection/fever).
* Caregiver Characteristics:

  * Has a child experiencing current acute complication of sickle cell disease, such as pain crisis, acute chest syndrome, stroke, or infection.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with sickle cell disease and their parents/guardians
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Descriptive group characteristics of sickle cell disease participants with and without nocturnal enuresis | Once at or near enrollment
  Health-related quality of life, emotional and behavioral functioning, family functioning, stressful life events, sociodemographic factors and medical factors will be examined from questionnaire responses. Classification will be based on the criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, text revision (DSM-IV-TR). Data will be stratified by age (6-11 years and 12-18 years) and genotype (HbSS/ HbSβ0 thalassemia and HbSC/ HbSβ+ thalassemia). The sample will be dichotomized using the binary response (by nocturnal enuresis/no nocturnal enuresis). Pearson's chi-square or Fisher's Exact test for categorical data and the two-sample t-test for continuous data will be performed to examine the group differences. Logistic regression will be performed using the binary response to examine the effect of these factors with covariates selected by Bayesian information criterion (BIC) with age group indicator and genotype included in the regression.

SECONDARY OUTCOMES:
Frequency of behavioral interventions | Once at or near enrollment
  The total number of interventions used and the frequencies of the type interventions used will be calculated. A summary will also be prepared for each age group (6-11 years and 12-18 years).
Barriers to the use of interventions to prevent nocturnal enuresis | Once at or near enrollment
  The number and frequencies of barriers to implementation of interventions will be assessed by a checklist of items (i.e., time, inconvenience, forgetfulness) and open-ended responses provided by participants. A summary will also be prepared for each age group (6-11 years and 12-18 years).

CONTACTS AND LOCATIONS:
Overall Officials: Jerlym Porter, PhD, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols